CLINICAL TRIAL: NCT05790369
Title: Effects of Home-Based Ankle Training Program on The Muscle Strength, Balance and Gait Function in the Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Principal Investigator, Hsiu-Chen Lin, Associate Professor, China Medical University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CMUH110-REC2-192
Record Dates: First submitted 2022-10-20; First posted 2023-03-30 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Aging
Keywords: Ankle strengthening training; Muscular strength; Balance ability; Gait function; Elderly
MeSH Terms: interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- New ankle machine training group (NAMTG) (Experimental): home-based ankle training program consisted of 6 exercises for their general physical fitness and use a device (new ankle machine) to provide progressive resisted exercise for the ankle strength
  Interventions: Behavioral: Resistance training (New ankle machine training)
- Elastic band training group (EBTG) (Active Comparator): home-based ankle training program consisted of 6 exercises for their general physical fitness and use Thera band to provide progressive resisted exercise for the ankle strength
  Interventions: Behavioral: Resistance training (Elastic band training )

INTERVENTIONS:
Behavioral: Resistance training (New ankle machine training) — A six week workout plan, the subjects receive on site or online guidance from professional coaches every two weeks.
  Arms: New ankle machine training group (NAMTG)
Behavioral: Resistance training (Elastic band training ) — A six week workout plan, the subjects receive on site or online guidance from professional coaches every two weeks.
  Arms: Elastic band training group (EBTG)

SUMMARY:
The occurrence of frequent falls influences the independence of the elderly's physical functions, and the factors related to falls include: weakness in the lower limbs, age, past injury experiences and so forth. Prolonged inactivity also increases the risk of falls, which is subsequently prone to bringing about other complications, which enhances the odds of falling again on the elderly.

In the literature, training methods for the lower limbs were for the most part of complex training, whereas only a few studied on the single part training. In locomotion, the ankle first touches the ground, needing strong ankle muscular strength to support the body. Nevertheless, previous studies rarely mentioned whether a single ankle muscular strength could reduce the risk of falls.

Traditionally, the training of ankle muscular strength practically utilizes elastic bands, and there are plenty of benefits confirmed in the literature. However, it is even harder to implement the operation in reality, especially in the elderly. To resolve this problem effectively, a new type of ankle training machine is added to this study. It can be adjusted to different levels of resistance, provide multi directional training, and allow the subjects to be trained in a sitting position achieving a stable state. In addition, this machine is easy to operate for the elderly.

The aims of this research are: (1) to propose two different types of ankle training methods and designed a 6 week training programs, (2) to explore whether the training programs can improve muscular strength, balance capacity and gait function and (3) compare the training effects between the two types of ankle training methods. In this study, 60 voluntary old citizens, aged over 65, will be recruited, and they will be randomly divided into: 30 members in the Elastic Band Training Group (EBTG) and 30 members in the New Ankle Training Machine Training Group (NAMTG). During the six week workout plan, the subjects receive on site or online guidance from professional coaches every two weeks; meanwhile, coaches can affirm whether the plan is executed properly, confirming the effectiveness of the home training. Through these two groups of home ankle training programs with different interventional approaches lasting six weeks, the objective of the intervention is to boost muscular strength, balance ability as well as gait ability, meanwhile to decline the risk of falls and to reduce high medical expenses and care labor costs.

ELIGIBILITY:
Inclusion Criteria:

* Healthy elderly people over 65 years old have no exercise habits.
* The ability to walk independently or without equipment is at least 10m.
* Able to independently perform activities related to daily life, such as doing housework, walking, climbing stairs, etc.
* Elderly people who have a history of minor stroke or upper limb surgery but have not affected the ankle movement can be included in the scope of the case.

Exclusion Criteria:

* There is a musculoskeletal system disease, or the movement of the limbs is severely restricted.
* If there is a history of lower limb surgery, which affects neurological symptoms and mobility, it is excluded.
* Exclude specific diseases, such as stroke, spinal cord injury,etc., who have obvious sequelae of movement.
* Participated in other programs including Muscular strength, Balance ability, Gait function training, etc. in the past 6 months

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 43 (Actual)
Dates: Start 2021-12-09 (Actual); Primary Completion 2023-01-08 (Actual); Study Completion 2023-01-08 (Actual)

PRIMARY OUTCOMES:
Muscle strength test | Change from Baseline (before the training) at the completion of 6 weeks training
  Sit-to-stand test, recoding by the time in seconds
Postural stability test | Change from Baseline (before the training) at the completion of 6 weeks training
  One-leg standing with eye-open and eye-closed, recoding by the the center of pressure from a force plate
Y- balance test | Change from Baseline (before the training) at the completion of 6 weeks training
  Recoding the distance in the anterior, posterio-medial and posterio-lateral in cm.
Gait analysis | Change from Baseline (before the training) at the completion of 6 weeks training
  Recoding the joint angle in degrees by the IMU sensors.

CONTACTS AND LOCATIONS:
Locations (1):
- China Medical University, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No